CLINICAL TRIAL: NCT04520178
Title: Effects of the Serotonin Precursor, 5-hydroxytryptophan, in the Injured Human Spinal Cord
Brief Title: Effects of 5HTP on the Injured Human Spinal Cord
Acronym: 5-HTP only
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Wings for Life (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00119483/00125176
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — 5-Hydroxytryptophan; Carbidopa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low-dose 5HTP (Active Comparator): 50mg 5-HTP in combination with 50mg carbidopa
  Interventions: Drug: 5-Hydroxytryptophan; Drug: Carbidopa
- High-dose 5HTP (Active Comparator): 100mg 5-HTP in combination with 50mg carbidopa
  Interventions: Drug: 5-Hydroxytryptophan 100 MG; Drug: Carbidopa
- Carbidopa (Sham Comparator): 50mg carbidopa only
  Interventions: Drug: Carbidopa
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5-Hydroxytryptophan 100 MG — 100mg combined with 50mg carbidopa
  Arms: High-dose 5HTP
Drug: 5-Hydroxytryptophan — 50mg combined with 50mg carbidopa
  Arms: Low-dose 5HTP
Drug: Carbidopa — 50mg
  Arms: Carbidopa; High-dose 5HTP; Low-dose 5HTP
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will assess how the serotonin precursor, 5-HTP, alter nervous system excitability and motor function in individuals with spinal cord injuries of differing chronicity and severity. Participants will visit the lab on 4 separate occasions where they will be administered four different drugs in a randomized, double-blinded, placebo-controlled crossover design.

DETAILED DESCRIPTION:
This study will assess for the first time the effects of 5-HTP on neural excitability utilizing a combination of neurophysiological and functional testing in subacute motor complete (AIS A/B), chronic motor complete (AIS A/B) and chronic incomplete (AIS C/D) SCI participants. To reduce peripheral side effects such as nausea, these supplements will be co-administered with carbidopa which inhibits the action of peripheral AADC, thereby ensuring that 5-HTP can effectively cross the blood brain barrier prior to being broken down. The neurophysiological outcomes will allow for the determination of the mechanistic actions of each pharmacological agent on different pathways/sites within the central nervous system in three different patient populations with varying degrees of lesion severity and will for the determination of whether increased Amino Acid Decarboxylase (AADC) expression and therefore the efficacy of this approach is correlated to lesion severity and/or chronicity. Importantly, the use of functional testing will allow for the determination of whether these often-reported neurophysiological changes translate to improvements in muscle activation patterns and kinematics during cycling.

The effects of 5-HTP will be assessed across three different participant groups: i) subacute (6 months-1 year) AIS A/B SCI individuals, ii) chronic (>2 years post injury) AIS A/B SCI individuals and iii) chronic AIS C/D SCI individuals.. In a placebo-controlled, randomized crossover design, participants will receive i) 50 mg 5HTP combined with 50 mg carbidopa, ii) 100 mg 5-HTP combined with 50 mg carbidopa, iii) 50 mg carbidopa only or iv) placebo. Ten participants will be recruited in each group. Participants will visit the lab on four separate occasions, separated by at least 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* participants must have suffered trauma to the spinal cord at least six months ago or longer

Exclusion Criteria:

* individuals with damage to the nervous system other than to the spinal cord
* pregnant and/or breastfeeding women
* alcoholic participants
* history of seizure/epilepsy
* history of suicidal thoughts or behaviors
* known or suspected allergy to the medication ingredients
* cardiovascular disease including history of heart attack or heart rhythm irregularities
* coronary artery disease
* reduced liver function or disease
* reduced kidney function or disease
* lung disease
* comatose or depressed states due to CNS depressants
* endocrine dysfunction
* blood dyscrasias or blood related disease
* bone marrow depression
* hypocalcemia
* history of stomach ulcers
* wide angle glaucoma
* phenylketonuria
* history of tumors
* uncontrolled heart problems
* unstable psychiatric or mental disorder

Participants taking:

* monoamine oxidase inhibitor therapy
* serotonergic antidepressants
* tricyclic antidepressants
* any type of serotonergic agonist
* dopamine D2 receptor antagonists
* amphetamine
* CNS depressants
* levodopa
* lithium
* anti-hypertensive drugs
* iron salts
* metoclopramide
* phenothiazine medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in motoneuron excitability | Pre drug-intake, 30minutes, 60minutes, 90minutes and 120minutes post drug-intake
  F waves
Change in spinal excitability | Pre drug-intake, 30minutes, 60minutes, 90minutes and 120minutes post drug-intake
  H reflex
Change in flexor reflex/spasms | Pre drug-intake, 30minutes, 60minutes, 90minutes and 120minutes post drug-intake
  Cutaneomuscular reflex
Change in functional movement performance | Pre drug-intake, 120-150minutes post drug-intake
  Leg cycling task

SECONDARY OUTCOMES:
Serum analysis of 5HIAA (UofL Cohort only) | 90-120minutes post drug-intake
  5-HIAA (serum)
Serum analysis of serotonin (UofL Cohort only) | 90-120minutes post drug-intake
  5-HT (serum and whole blood), cortisol
Serum analysis of cortisol (UofL Cohort only) | 90-120minutes post drug-intake
  serum cortisol
Whole blood analysis of Serotonin (UofL Cohort only) | 90-120minutes post drug-intake
  Blood 5HT

CONTACTS AND LOCATIONS:
Overall Officials: Jessica D'Amico, PhD, Principal Investigator — University of Alberta
Locations (2):
- University of Louisville, Louisville, Kentucky, United States
- University of Alberta, Edmonton, Alberta, Canada